CLINICAL TRIAL: NCT04879732
Title: Roentgen Stereophotogrammetric Analysis (RSA): ACTIS Hip Stem
Brief Title: RSA - ACTIS Hip Stem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Radiostereometric Analysis Network (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B2021:005
Record Dates: First submitted 2021-04-30; First posted 2021-05-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ACTIS hip stem (Other): All participants will receive the ACTIS hip stem.
  Interventions: Device: ACTIS

INTERVENTIONS:
Device: ACTIS — ACTIS Hip stem

SUMMARY:
The principal objective of this study is to compare mean 2-year subsidence of the ACTIS femoral stem using model-based RSA against published migration patterns for hip stems of a similar design. Secondary objectives include comparison of migration per surgical approach, quantifying changes in functional and health status of subjects following surgery, and assess occurrences of complications and adverse events.

DETAILED DESCRIPTION:
This is a multi-centre, sequential enrollment trial of patients undergoing primary total hip arthroplasty. Patients will be recruited at three Canadian Centres to receive the ACTIS femoral hip stem via 3 different surgical approaches.

Model-based RSA will identify migration of the implant with respect to the femoral bone during the first 2 post-operative years. Patient health and functional outcomes will be recorded at pre- and post-operative intervals to quantify improvement as a result of the surgery and trajectory of recovery. Adverse events and clinical complications in each study group will be captured and compared. Select surgical, hospital and rehabilitation data will be collected to measure health economic outcomes relating to the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the hip indicating primary total hip arthroplasty
* Aged 21 years or older
* Patients willing and able to comply with follow-up requirements and self-evaluations
* Ability to give informed consent
* Body mass index ≤45 kg/m2

Exclusion Criteria

* Active or prior infection
* Medical condition precluding major surgery
* Medical condition with less than 2 years life expectancy
* Overhanging pannus (for anterior approach cohort only)
* Prior surgery of the hip involving implantation of hardware (i.e., hemiarthroplasty, internal fixation, pelvic reconstruction near the acetabulum requiring removal)
* Skin condition on the area of incision
* Multi-level lumbar spine fusion
* Ankylosing spondylolithesis
* Shortening osteotomy through the femur

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Subsidence of the ACTIS femoral stem | 2 Year
  Compare mean 2-year subsidence using model-based RSA (radiostereometric analysis) (mm). The images taken at each time point will be compared with the baseline to assess the change in implant position.

SECONDARY OUTCOMES:
Comparison of migration per surgical approach | 2 Year
  Comparison between the 3 approaches (postero-lateral, direct lateral, and direct anterior); measured migration (mm). The images taken at each time point will be compared with the baseline to assess implant migration. Therefore the outcome is change in implant position measured using RSA.
Oxford Hip Score (OHS) | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in functional outcomes assessments, patient reported outcome. Each item is scored from 0 to 4, and the items are summated, with lower total scores indicating poorer performance.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups and timepoints. The scores in each section (pain, stiffness and function limitation) are totaled; 5 items for pain (score range 0-20), 2 for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
European Quality of Life (EQ-5D-5L) questionnaire | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in functional outcomes assessments, patient reported outcome. A health state score is obtained based on the responses from 1-5 in each subscale, from which a single index value is calculated representing patients' overall health state. The overall health state range from 0 to 1.0.
Visual analogue scale (VAS) for thigh pain | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported satisfaction as measured using the visual analogue scale (VAS) from 0 (No pain) - 100 (Worst pain imaginable).
Visual analogue scale (VAS) for satisfaction | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change from preoperative to 2 years between the study groups timepoints in patient reported pain severity as measured using the visual analogue scale (VAS) from 0 (Unsatisfied) - 100 (Completely satisfied).
University of California at Los Angeles (UCLA) Activity Level scale | Preoperative, 6 Weeks, 3 Months, 6 Months, 1 Year and 2 Years
  Evaluate and compare the change in UCLA activity score compared to baseline in the study cohort. UCLA activity scores range from 1 to 10, and is a measure of activity with 10 being most active.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Turgeon, MD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - Orthopaedic Innovation Centre, Winnipeg, Manitoba
  - Nova Scotia Health - Orthopedic, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol